CLINICAL TRIAL: NCT06368193
Title: The Neuralert Stroke Monitor Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralert Technologies LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Neuralert 001
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Surgery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cardiac Surgery Patients OR Neurology Patients (Experimental)
  Interventions: Device: Neuralert Monitor

INTERVENTIONS:
Device: Neuralert Monitor — Device to identify upper extremity asymmetry in patients who are high risk for stroke.

SUMMARY:
This trial aims to demonstrate that the Neuralert Monitoring System will detect strokes before they would be identified by current standard of care. Each patient will be monitored for up to five days, depending on device connectivity or battery duration. Each monitoring session will consist of wearing a Neuralert device on each arm. For this pilot trial, we are interested in learning about Wi-Fi connectivity, successful data transmission, integration into clinical workflow, usability and tolerability.

ELIGIBILITY:
1. Male or female age ≥ 22 years
2. Admitted or planned admission to one of the participating hospitals and followed by the Cardiothoracic (CT) Surgery or Vascular Surgery services
3. Considered at high risk for stroke while in the hospital based on:

   Ø Interventions or procedures that are high-risk for stroke performed during the hospitalization, which may include:
   * Intracardiac surgical or endovascular procedures, including valve replacement
   * Ascending aorta or aortic arch surgical or endovascular repair
   * Open surgical or endovascular carotid revascularization

   Ø Other cardiac procedures along with a high-risk medical history:
   * Age ≥ 80 years · Prior stroke/TIA
   * Hypercoagulable state (i.e., prior clotting events attributed to active malignancy or a diagnosed thrombophilia) requiring lifelong anticoagulation
   * Severely reduced left ventricular cardiac ejection fraction (i.e., <30%) or anterior left ventricular wall akinesis
   * Atrial fibrillation
4. Admitted with a stroke or TIA attributed to large artery occlusion or severe stenosis that has not been revascularized.

Exclusion Criteria: (all must be no)

1. Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
2. Baseline preoperative asymmetric upper extremity weakness as assessed by the Investigator, defined as a differential in the NIHSS upper extremity motor score between the two arms of >0
3. Above the wrist amputation
4. Unwilling to provide informed consent or no legally authorized representative willing to provide consent if the patient is unable
5. Currently imprisoned

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to Nursing Response | Up to 5 days post patient surgery
  The time from the nurse receiving an alert to the time they respond after assessing the patient.
Time to Generate Alert | Up to 5 days post patient surgery
  The time to successful generation of an alert to staff when asymmetry or low battery is detected.

SECONDARY OUTCOMES:
Number of Strokes Identified | Up to 5 days post patient surgery
  The number of strokes identified by the Neuralert device and the number of strokes identified by usual care. If a stroke is identified at the next clinical evaluation after an alarm occurs, it will be considered to have been detected by the Neuralert device.
Device Tolerability | Up to 5 days post patient surgery
  The tolerability and impact on clinical workflow and patient feedback on tolerability after study completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Messe SR, Kasner SE, Cucchiara BL, McGarvey ML, Cummings S, Acker MA, Desai N, Atluri P, Wang GJ, Jackson BM, Weimer J. Derivation and Validation of an Algorithm to Detect Stroke Using Arm Accelerometry Data. J Am Heart Assoc. 2023 Feb 7;12(3):e028819. doi: 10.1161/JAHA.122.028819. Epub 2023 Jan 31. PMID 36718858